CLINICAL TRIAL: NCT00937937
Title: A Phase II Trial of SCH 727965 (NSC 747135) in Patients With Stage IV Melanoma
Brief Title: Dinaciclib in Treating Patients With Stage IV Melanoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2011-01935; NCI-2011-01935 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); SWOG-S0826; CDR0000647155; S0826 (Other: SWOG); S0826 (Other: CTEP); U10CA032102 (NIH)
Record Dates: First submitted 2009-07-10; First posted 2009-07-13 (Estimated); Results first posted 2016-07-22 (Estimated); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Acral Lentiginous Melanoma; Cutaneous Nodular Melanoma; Lentigo Maligna Melanoma; Low-CSD Melanoma; Mucosal Melanoma; Recurrent Melanoma; Stage IV Cutaneous Melanoma AJCC v6 and v7
MeSH Terms: conditions — Melanoma | interventions — dinaciclib

ARMS (1):
- Arm I (Experimental): Patients receive dinaciclib IV over 2 hours on day 1. Treatment repeats every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Dinaciclib

INTERVENTIONS:
Drug: Dinaciclib — Given IV
  Other Names: CDK Inhibitor SCH 727965; MK 7965; MK-7965; MK7965; SCH 727965; SCH-727965; SCH727965

SUMMARY:
This phase II trial is studying the side effects and how well dinaciclib works in treating patients with stage IV melanoma. Dinaciclib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the 1-year overall survival rate in patients with stage IV melanoma treated with dinaciclib.

SECONDARY OBJECTIVES:

I. To assess the 6-month progression-free survival rate in these patients. II. To evaluate the response rate (confirmed and unconfirmed complete and partial responses) in the subset of patients with measurable disease.

III. To assess the safety and tolerability of dinaciclib given to patients with stage IV melanoma.

OUTLINE: This is a multicenter study.

Patients receive dinaciclib IV over 2 hours on day 1. Treatment repeats every 21 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 6 months for up to 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy-confirmed malignant melanoma

  * Stage IV disease
  * Cutaneous or mucosal origin
  * Melanoma of unknown primary allowed
  * No ocular melanoma
* Measurable or non-measurable disease
* No prior or concurrent brain metastases as confirmed by CT scan or MRI
* Zubrod performance status 0-1
* ANC ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Hemoglobin ≥ 9 g/dL
* Serum bilirubin ≤ 1.5 times upper limit of normal (ULN) (including patients with hepatic metastases)
* SGOT or SGPT ≤ 2.5 times ULN (≤ 5 times ULN in the presence of hepatic metastases)
* Serum creatinine ≤ 1.5 times ULN
* Not pregnant or nursing
* Fertile patients must use effective contraception
* No other prior malignancy except for adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, adequately treated stage I or II cancer from which the patient is currently in complete remission, or any other cancer from which the patient has been disease-free for 5 years
* No prior therapy with a cyclin-dependent kinase inhibitor
* At least 14 days since prior radiotherapy
* At least 28 days since prior systemic chemotherapy
* At least 28 days since prior adjuvant systemic therapy
* At least 28 days since prior surgery
* No more than 1 prior systemic therapy regimen (chemotherapy, biologic/immunotherapy, hormonal therapy, or a combination regimen) for stage IV melanoma and any side effects must have resolved to ≤ grade 1
* Any number of prior adjuvant systemic therapy regimens allowed, including interferon alfa-2b, GM-CSF, chemotherapy, and chemobiotherapy

  * Therapy for stage IV resected free-of-disease will be considered adjuvant therapy
* Prior radiotherapy allowed provided any side effects have resolved to ≤ grade 1
* Prior surgery (for both the primary and stage IV disease) allowed provided side effects have resolved to ≤ grade 1
* No other concurrent or planned non-study treatment (including chemotherapy, hormonal therapy, biologic therapy, or radiotherapy)
* No concurrent CYP3A4 inhibitors or inducers
* No concurrent grapefruit or grapefruit juice

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2009-07-01 (Actual); Primary Completion 2013-10-22 (Actual); Study Completion 2026-03-19 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher D Lao, Principal Investigator — SWOG Cancer Research Network
Locations (190):
- United States (190):
  - Providence Hospital, Mobile, Alabama
  - Mercy Hospital Fort Smith, Fort Smith, Arkansas
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Highlands Oncology Group - Rogers, Rogers, Arkansas
  - East Bay Radiation Oncology Center, Castro Valley, California
  - Eden Hospital Medical Center, Castro Valley, California
  - Valley Medical Oncology Consultants-Castro Valley, Castro Valley, California
  - Bay Area Breast Surgeons Inc, Emeryville, California
  - Valley Medical Oncology Consultants-Fremont, Fremont, California
  - Contra Costa Regional Medical Center, Martinez, California
  - El Camino Hospital, Mountain View, California
  - Wilma Chan Highland Hospital, Oakland, California
  - Alta Bates Summit Medical Center - Summit Campus, Oakland, California
  - Bay Area Tumor Institute, Oakland, California
  - Hematology and Oncology Associates-Oakland, Oakland, California
  - Tom K Lee Inc, Oakland, California
  - UC Irvine Health/Chao Family Comprehensive Cancer Center, Orange, California
  - Valley Care Health System - Pleasanton, Pleasanton, California
  - Valley Medical Oncology Consultants, Pleasanton, California
  - Doctors Medical Center- JC Robinson Regional Cancer Center, San Pablo, California
  - Poudre Valley Hospital, Fort Collins, Colorado
  - Smilow Cancer Hospital Care Center at Saint Francis, Hartford, Connecticut
  - Boca Raton Comprehensive Cancer Center, Boca Raton, Florida
  - Orlando Health Cancer Institute, Orlando, Florida
  - Memorial Health University Medical Center, Savannah, Georgia
  - Lewis Cancer and Research Pavilion at Saint Joseph's/Candler, Savannah, Georgia
  - South Georgia Medical Center/Pearlman Cancer Center, Valdosta, Georgia
  - OSF Saint Anthony's Health Center, Alton, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Advocate Good Samaritan Hospital, Downers Grove, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - SSM Health Good Samaritan, Mount Vernon, Illinois
  - Springfield Memorial Hospital, Springfield, Illinois
  - Franciscan Saint Francis Health-Beech Grove, Beech Grove, Indiana
  - Reid Health, Richmond, Indiana
  - Cancer Center of Kansas - Chanute, Chanute, Kansas
  - Cancer Center of Kansas - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - HaysMed, Hays, Kansas
  - Hutchinson Regional Medical Center, Hutchinson, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - University of Kansas Cancer Center, Kansas City, Kansas
  - Cancer Center of Kansas-Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Southwest Medical Center, Liberal, Kansas
  - Cancer Center of Kansas-Liberal, Liberal, Kansas
  - Cancer Center of Kansas - Newton, Newton, Kansas
  - Olathe Cancer Center, Olathe, Kansas
  - Menorah Medical Center, Overland Park, Kansas
  - Saint Luke's South Hospital, Overland Park, Kansas
  - Cancer Center of Kansas - Parsons, Parsons, Kansas
  - Mercy Hospital Pittsburg, Pittsburg, Kansas
  - Kansas City NCI Community Oncology Research Program, Prairie Village, Kansas
  - Cancer Center of Kansas - Pratt, Pratt, Kansas
  - Cancer Center of Kansas - Salina, Salina, Kansas
  - Salina Regional Health Center, Salina, Kansas
  - AdventHealth Shawnee Mission, Shawnee Mission, Kansas
  - Cotton O'Neil Cancer Center / Stormont Vail Health, Topeka, Kansas
  - University of Kansas Health System Saint Francis Campus, Topeka, Kansas
  - Cancer Center of Kansas - Wellington, Wellington, Kansas
  - Associates In Womens Health, Wichita, Kansas
  - Cancer Center of Kansas-Wichita Medical Arts Tower, Wichita, Kansas
  - Ascension Via Christi Hospitals Wichita, Wichita, Kansas
  - Cancer Center of Kansas - Wichita, Wichita, Kansas
  - Wichita NCI Community Oncology Research Program, Wichita, Kansas
  - Cancer Center of Kansas - Winfield, Winfield, Kansas
  - Baton Rouge General Medical Center, Baton Rouge, Louisiana
  - Mary Bird Perkins Cancer Center, Baton Rouge, Louisiana
  - Louisiana State University Health Science Center, New Orleans, Louisiana
  - University Medical Center New Orleans, New Orleans, Louisiana
  - Boston Medical Center, Boston, Massachusetts
  - Michigan Cancer Research Consortium NCORP, Ann Arbor, Michigan
  - Trinity Health Saint Joseph Mercy Hospital Ann Arbor, Ann Arbor, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Bronson Battle Creek, Battle Creek, Michigan
  - Spectrum Health Big Rapids Hospital, Big Rapids, Michigan
  - Corewell Health Dearborn Hospital, Dearborn, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Health Saint John Hospital, Detroit, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Genesys Regional Medical Center-West Flint Campus, Flint, Michigan
  - Cancer Research Consortium of West Michigan NCORP, Grand Rapids, Michigan
  - Corewell Health Grand Rapids Hospitals - Butterworth Hospital, Grand Rapids, Michigan
  - Trinity Health Grand Rapids Hospital, Grand Rapids, Michigan
  - Allegiance Health, Jackson, Michigan
  - University of Michigan Health - Sparrow Lansing, Lansing, Michigan
  - Trinity Health Saint Mary Mercy Livonia Hospital, Livonia, Michigan
  - Trinity Health Muskegon Hospital, Muskegon, Michigan
  - Trinity Health Saint Joseph Mercy Oakland Hospital, Pontiac, Michigan
  - Lake Huron Medical Center, Port Huron, Michigan
  - MyMichigan Medical Center Saginaw, Saginaw, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Henry Ford Health Warren Hospital, Warren, Michigan
  - University of Michigan Health - West, Wyoming, Michigan
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - University Health Truman Medical Center, Kansas City, Missouri
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - Saint Joseph Health Center, Kansas City, Missouri
  - North Kansas City Hospital, Kansas City, Missouri
  - Heartland Hematology and Oncology Associates Incorporated, Kansas City, Missouri
  - Research Medical Center, Kansas City, Missouri
  - Saint Luke's East - Lee's Summit, Lee's Summit, Missouri
  - Liberty Hospital, Liberty, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Mercy Infusion Center - Chippewa, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Saint Louis-Cape Girardeau CCOP, St Louis, Missouri
  - Billings Clinic Cancer Center, Billings, Montana
  - Northern Rockies Radiation Oncology Center, Billings, Montana
  - Saint Vincent Healthcare, Billings, Montana
  - Montana Cancer Consortium NCORP, Billings, Montana
  - Saint Vincent Frontier Cancer Center, Billings, Montana
  - Bozeman Health Deaconess Hospital, Bozeman, Montana
  - Saint James Community Hospital and Cancer Treatment Center, Butte, Montana
  - Benefis Sletten Cancer Institute, Great Falls, Montana
  - Berdeaux, Donald MD (UIA Investigator), Great Falls, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Northern Montana Hospital, Havre, Montana
  - Saint Peter's Community Hospital, Helena, Montana
  - Glacier Oncology PLLC, Kalispell, Montana
  - Kalispell Medical Oncology, Kalispell, Montana
  - Logan Health Medical Center, Kalispell, Montana
  - Montana Cancer Specialists, Missoula, Montana
  - Saint Patrick Hospital - Community Hospital, Missoula, Montana
  - Community Medical Center, Missoula, Montana
  - Guardian Oncology and Center for Wellness, Missoula, Montana
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - Nevada Cancer Institute-Summerlin Campus, Las Vegas, Nevada
  - University of Rochester, Rochester, New York
  - Novant Health Presbyterian Medical Center, Charlotte, North Carolina
  - Wayne Memorial Hospital, Goldsboro, North Carolina
  - FirstHealth of the Carolinas-Moore Regional Hospital, Pinehurst, North Carolina
  - Southeast Clinical Oncology Research Consortium NCORP, Winston-Salem, North Carolina
  - Grandview Hospital, Dayton, Ohio
  - Good Samaritan Hospital - Dayton, Dayton, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Miami Valley Hospital North, Dayton, Ohio
  - Dayton NCI Community Oncology Research Program, Dayton, Ohio
  - Blanchard Valley Hospital, Findlay, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - Clinton Memorial Hospital/Foster J Boyd Regional Cancer Center, Wilmington, Ohio
  - Greene Memorial Hospital, Xenia, Ohio
  - Saint Charles Health System, Bend, Oregon
  - Providence Milwaukie Hospital, Milwaukie, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Adventist Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Salem Hospital, Salem, Oregon
  - Prisma Health Cancer Institute - Spartanburg, Boiling Springs, South Carolina
  - Prisma Health Cancer Institute - Easley, Easley, South Carolina
  - McLeod Regional Medical Center, Florence, South Carolina
  - Greenville Health System Cancer Institute-Andrews, Greenville, South Carolina
  - Saint Francis Hospital, Greenville, South Carolina
  - Prisma Health Cancer Institute - Butternut, Greenville, South Carolina
  - Prisma Health Cancer Institute - Faris, Greenville, South Carolina
  - Prisma Health Greenville Memorial Hospital, Greenville, South Carolina
  - Prisma Health Cancer Institute - Eastside, Greenville, South Carolina
  - Self Regional Healthcare, Greenwood, South Carolina
  - Prisma Health Cancer Institute - Greer, Greer, South Carolina
  - Prisma Health Cancer Institute - Seneca, Seneca, South Carolina
  - Wellmont Holston Valley Hospital and Medical Center, Kingsport, Tennessee
  - Thompson Cancer Survival Center, Knoxville, Tennessee
  - Medical City Dallas Hospital, Dallas, Texas
  - Scott and White Memorial Hospital, Temple, Texas
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - Danville Regional Medical Center, Danville, Virginia
  - Sovah Health Martinsville, Martinsville, Virginia
  - Ballad Health Cancer Care - Norton, Norton, Virginia
  - PeaceHealth Saint Joseph Medical Center, Bellingham, Washington
  - Kadlec Clinic Hematology and Oncology, Kennewick, Washington
  - Skagit Valley Hospital, Mount Vernon, Washington
  - Harrison HealthPartners Hematology and Oncology-Poulsbo, Poulsbo, Washington
  - Harborview Medical Center, Seattle, Washington
  - Minor and James Medical PLLC, Seattle, Washington
  - Fred Hutchinson Cancer Center, Seattle, Washington
  - Kaiser Permanente Washington, Seattle, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - University of Washington Medical Center - Montlake, Seattle, Washington
  - Saint Michael Cancer Center, Silverdale, Washington
  - Cancer Care Northwest - Spokane South, Spokane, Washington
  - Evergreen Hematology and Oncology PS, Spokane, Washington
  - PeaceHealth Southwest Medical Center, Vancouver, Washington
  - Wenatchee Valley Hospital and Clinics, Wenatchee, Washington
  - Rocky Mountain Oncology, Casper, Wyoming
  - Welch Cancer Center, Sheridan, Wyoming

REFERENCES:
- [Derived] Lao CD, Moon J, Ma VT, Fruehauf JP, Flaherty LE, Bury MJ, Martin WG, Gross H, Akerley W, Hopkins JO, Patel SP, Sondak VK, Ribas A. Southwest Oncology Group S0826: A phase 2 trial of SCH 727965 (NSC 727135, dinaciclib) in patients with stage IV melanoma. Cancer. 2025 Jan 1;131(1):e35587. doi: 10.1002/cncr.35587. Epub 2024 Sep 29. PMID 39342463

RESULTS

PARTICIPANT FLOW:
Groups:
- Dinaciclib: Patients receive dinaciclib IV over 2 hours on day 1. Treatment repeats every 21 days in the absence of disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Dinaciclib
Started | 72
Completed | 0
Not Completed | 72
Not completed — Adverse Event | 6
Not completed — Withdrawal by Subject | 2
Not completed — Progression/relapse | 61
Not completed — Death | 1
Not completed — Other | 2

BASELINE CHARACTERISTICS:
Population: Include all the patients that have received the treatment and been adverse event evaluable.
Arm/Group | Dinaciclib
Number analyzed (Participants) | 72
Age, Continuous [Median (Full Range); unit: years] — The median ans full range of those 72 patients' ages.
  years | 65.4 [28.6 to 90.4]
Sex: Female, Male [Count of Participants; unit: Participants] — The gender summary of those 72 patients who have received Dinaciclib.
  Participants
    Female | 20
    Male | 52
Race/Ethnicity, Customized [Number; unit: participants] — The race summary of 72 patients who have received Dinaciclib.
  participants
    White | 69
    Asian | 2
    Pacific Islander | 1
Hispanic [Number; unit: participants] — The hispanic or non-hispanic summary of 72 patients who have received Dinaciclib.
  participants
    Yes | 2
    No | 69
    Unknown | 1
Performance Status [Number; unit: participants] — The performance status of 72 patients who have received Dinaciclib. Only performance status 0 or 1 are included in the study.
  Performance status 0: Fully active, able to carry on all pre-disease performance without restriction.
  Performance status 1: Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work.
  The higher score, the worse outcomes.
  participants
    0 | 38
    1 | 34
Site(s) of Metastases [Number; unit: participants] — Sites of metastases of 72 patients who have received Dinaciclib.
  participants
    Bone | 18
    Brain | 0
    Liver | 23
    Lymph node, soft tissue, skin | 41
    Lung | 41
    Other visceral | 17
    Other non-visceral | 14
Elevated LDH [Number; unit: participants] — Whether elevated LDH or not of 72 patients who have received Dinaciclib.
  participants
    No | 41
    Yes | 31
Primary Type [Number; unit: participants] — Primary type of melanoma of 72 patients who have received Dinaciclib.
  participants
    Cutaneous | 55
    Mucosal | 8
    Unknown primary | 9

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: From date of registration to date of death due to any cause. Patients last known to be alive are censored at date of last contact.
Time Frame: Weekly, up to 3 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Dinaciclib
Number analyzed (Participants) | 72
months | 8 [6 to 11]
Statistical Analysis 1: Comparison: Dinaciclib; one-year overall survival estimate; Test type: Superiority or Other; 1-year overall survival estimate = 0.38, 95% CI 2-sided [0.27 to 0.49]

2. Secondary Outcome: Progression-free Survival Assessed by Response Evaluation Criteria for Solid Tumors (RECIST)
Description: Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions. The duration from the date of randomization to the date of first documentation of progressive disease, symptomatic deterioration, or death dure to any cause.
Time Frame: Disease assessment was performed every 6 weeks, up to 3 years.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Dinaciclib
Number analyzed (Participants) | 72
months | 1.4 [1.4 to 1.5]
Statistical Analysis 1: Comparison: Dinaciclib; 6-month PFS estimate; Test type: Superiority or Other; 6-month PFS estimate = 0.07, 95% CI 2-sided [0.03 to 0.15]

3. Secondary Outcome: Response Rate (Confirmed and Unconfirmed Complete and Partial Responses) Assessed by RECIST
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: Disease assessments for response were performed every 6 weeks, up to 3 years
Measure: Mean (95% Confidence Interval); unit: percentage of participants
Arm/Group | Dinaciclib
Number analyzed (Participants) | 72
percentage of participants | 0 [0 to 0.05]

4. Secondary Outcome: Number of Patients With Gr 3 Through 5 Adverse Events That Are Related to Study Drugs
Description: Adverse Events (AEs) are reported by CTCAE Version 3.0. Only adverse events that are possibly, probably or definitely related to study drug are reported. The outcome measure here is different from Serious Adverse Event, whose definition could be more strict and specific. The number of patients who suffers the certain adverse event listed here could be larger than the number listed in following serious adverse event.
Time Frame: Toxicity assessment was evaluated after each cycle (21 days), up to 3 years.
Population: Eligible patients who had received the protocol treatments were included in the adverse event summaries. Any CTCAE 3.0 event of Grade 3 (serious), Grade 4 (life threatening) or Grade 5 (fatal) which were deemed to be related to protocol treatment are included.
Measure: Number; unit: Participants
Arm/Group | Dinaciclib
Number analyzed (Participants) | 72
Participants
  AST, SGOT | 1
  Cardiac troponin I (cTnI) | 1
  Cardiac-ischemia/infarction | 1
  Constitutional Symptoms-Other (Specify) | 1
  Dehydration | 1
  Diarrhea | 11
  Dyspnea (shortness of breath) | 1
  Edema: limb | 1
  Fatigue (asthenia, lethargy, malaise) | 3
  Febrile neutropenia | 2
  Hypotension | 2
  Hypoxia | 1
  Leukocytes (total WBC) | 18
  Lymphopenia | 5
  Metabolic/Laboratory-Other (Specify) | 2
  Mucositis/stomatitis (clinical exam) - Oral cavity | 1
  Muscle weakness, not d/t neuropathy - body/general | 1
  Nausea | 1
  Neutrophils/granulocytes (ANC/AGC) | 36
  Ocular/Visual-Other (Specify) | 1
  PTT (Partial thromboplastin time) | 1
  Pain - Abdomen NOS | 2
  Pain - Back | 1
  Pain - Cardiac/heart | 1
  Pain - Extremity-limb | 1
  Pain - Head/headache | 1
  Pain - Tumor pain | 1
  Prolonged QTc interval | 1
  Renal failure | 1
  SVT and nodal arrhythmia - Atrial fibrillation | 1
  SVT and nodal arrhythmia - Atrial flutter | 1
  SVT and nodal arrhythmia - Sinus tachycardia | 1
  Sodium, serum-low (hyponatremia) | 1
  Somnolence/depressed level of consciousness | 1
  Syncope (fainting) | 1
  Thrombosis/thrombus/embolism | 1
  Vascular-Other (Specify) | 1
  Vision-blurred vision | 1
  Vomiting | 1

ADVERSE EVENTS:
Time Frame: Toxicity assessment was evaluated after each cycle (21 days), up to 3 years.
Arm/Group | SCH 727965
Serious Adverse Events (participants affected / at risk) | 30/72
Other Adverse Events (participants affected / at risk) | 64/72
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SCH 727965 (N=72)
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Hemoglobin (Blood and lymphatic system disorders) | 1
Pain - Cardiac/heart (Cardiac disorders) | 1
SVT and nodal arrhythmia - Atrial fibrillation (Cardiac disorders) | 2
Ocular/Visual-Other (Eye disorders) | 1
Vision-blurred vision (Eye disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1
Pain - Abdomen NOS (Gastrointestinal disorders) | 1
Death not associated with CTCAE term - Death NOS (General disorders) | 1
Edema: limb (General disorders) | 1
Edema: trunk/genital (General disorders) | 1
Pain - Chest/thorax NOS (General disorders) | 1
Pain-Other (General disorders) | 2
Fracture (Injury, poisoning and procedural complications) | 1
AST, SGOT (Investigations) | 1
Alkaline phosphatase (Investigations) | 1
Cardiac troponin I (cTnI) (Investigations) | 1
Leukocytes (total WBC) (Investigations) | 2
Lymphopenia (Investigations) | 1
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 13
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 3
Phosphate, serum-low (hypophosphatemia) (Metabolism and nutrition disorders) | 1
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 2
Muscle weakness, not d/t neuropathy - body/general (Musculoskeletal and connective tissue disorders) | 1
Pain - Back (Musculoskeletal and connective tissue disorders) | 1
Pain - Extremity-limb (Musculoskeletal and connective tissue disorders) | 1
Trismus (diff, restriction, pain opening mouth) (Musculoskeletal and connective tissue disorders) | 1
Death - Disease progression NOS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8
Pain - Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Neuropathy: motor (Nervous system disorders) | 1
Neuropathy: sensory (Nervous system disorders) | 1
Ocular/Visual-Other (Nervous system disorders) | 1
Pain - Head/headache (Nervous system disorders) | 1
Somnolence/depressed level of consciousness (Nervous system disorders) | 1
Syncope (fainting) (Nervous system disorders) | 1
Renal failure (Renal and urinary disorders) | 1
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 3
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 1
Hypotension (Vascular disorders) | 3
Thrombosis/thrombus/embolism (Vascular disorders) | 1
Vascular-Other (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | SCH 727965 (N=72)
Hemoglobin (Blood and lymphatic system disorders) | 30
Vision-blurred vision (Eye disorders) | 4
Constipation (Gastrointestinal disorders) | 18
Diarrhea (Gastrointestinal disorders) | 43
Heartburn/dyspepsia (Gastrointestinal disorders) | 4
Mucositis/stomatitis (clinical exam) - Oral cavity (Gastrointestinal disorders) | 5
Nausea (Gastrointestinal disorders) | 42
Pain - Abdomen NOS (Gastrointestinal disorders) | 10
Vomiting (Gastrointestinal disorders) | 30
Edema: limb (General disorders) | 8
Fatigue (asthenia, lethargy, malaise) (General disorders) | 45
Fever in absence of neutropenia, ANC lt1.0x10e9/L (General disorders) | 7
Rigors/chills (General disorders) | 7
Infection-Other (Infections and infestations) | 5
ALT, SGPT (serum glutamic pyruvic transaminase) (Investigations) | 9
AST, SGOT (Investigations) | 9
Alkaline phosphatase (Investigations) | 8
Bilirubin (hyperbilirubinemia) (Investigations) | 4
Creatinine (Investigations) | 9
Leukocytes (total WBC) (Investigations) | 40
Lymphopenia (Investigations) | 13
Metabolic/Laboratory-Other (Investigations) | 5
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 41
Platelets (Investigations) | 4
Weight loss (Investigations) | 4
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 12
Anorexia (Metabolism and nutrition disorders) | 16
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 8
Dehydration (Metabolism and nutrition disorders) | 5
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 14
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 6
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 8
Muscle weakness, not d/t neuropathy - body/general (Musculoskeletal and connective tissue disorders) | 4
Pain - Back (Musculoskeletal and connective tissue disorders) | 12
Pain - Extremity-limb (Musculoskeletal and connective tissue disorders) | 7
Pain - Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6
Dizziness (Nervous system disorders) | 5
Neuropathy: sensory (Nervous system disorders) | 4
Pain - Head/headache (Nervous system disorders) | 7
Taste alteration (dysgeusia) (Nervous system disorders) | 8
Mood alteration - depression (Psychiatric disorders) | 5
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 6
Cough (Respiratory, thoracic and mediastinal disorders) | 16
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 8
Dermatology/Skin-Other (Skin and subcutaneous tissue disorders) | 4
Hair loss/Alopecia (scalp or body) (Skin and subcutaneous tissue disorders) | 11
Rash/desquamation (Skin and subcutaneous tissue disorders) | 6
Sweating (diaphoresis) (Skin and subcutaneous tissue disorders) | 7
Hypotension (Vascular disorders) | 16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less